CLINICAL TRIAL: NCT05978609
Title: Efficacy and Safety of Cadonilimab Combined With Gemcitabine and Cisplatin in the First-line Treatment of Unresectable Locally Advanced or Metastatic Biliary Malignancies
Brief Title: Cadonilimab With Chemotherapy in Treating Advanced Biliary Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Wentao Wang, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1036
Record Dates: First submitted 2023-07-18; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Cholangiocarcinoma Non-resectable
MeSH Terms: interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Candonilimab in combination with cisplatin and gemcitabine (Experimental): This study is a single-arm study to evaluate the safety and efficacy of candonilimab combined with cisplatin and gemcitabine in advanced biliary tract tumors
  Candonilimab 10mg/kg, Ivgtt，Q3W，Every 21 days is a cycle, administered on the first day of each cycle, and used continuously；
  Cisplatin，25mg/m2，Ivgtt，Dosing on days 1 and 8，Every 21 days is a cycle, administered on the first day of each cycle, and used continuously；
  gemcitabine 1000mg/m2，Ivgtt，Dosing on days 1 and 8，Every 21 days is a cycle, administered on the first day of each cycle, and used continuously；
  Interventions: Drug: Candonilimab; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Candonilimab — Candonilimab 10mg/kg, Ivgtt，Q3W，Every 21 days is a cycle, administered on the first day of each cycle, and used continuously；
Drug: Cisplatin — Cisplatin，25mg/m2，Ivgtt，Dosing on days 1 and 8，Every 21 days is a cycle, administered on the first day of each cycle, and used continuously；
Drug: Gemcitabine — gemcitabine 1000mg/m2，Ivgtt，Dosing on days 1 and 8，Every 21 days is a cycle, administered on the first day of each cycle, and used continuously；

SUMMARY:
The goal of this single-arm, Phase II interventional clinical trial is to test the safety and effectiveness of a combination treatment using the Cadonilimab with Gemcitabine and Cisplatin in patients with unresectable, locally advanced or metastatic biliary tract malignancies. The main questions it aims to answer are:

* Is this combined treatment protocol safe for these patients?
* Is this combined treatment protocol effective in treating these patients?

Participants will be given a combination treatment of Cadonilimab, Gemcitabine, and Cisplatin. Researchers will monitor their health conditions to assess the safety and effectiveness of this treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain written informed consent before implementing any experimental procedures.
2. Age between 18 and 75 years (any gender).
3. Histologically or cytologically confirmed unresectable locally advanced or metastatic biliary tumors (intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder carcinoma).
4. No prior systemic treatment, curative surgery, or adjuvant therapy allowed within the past 6 months.
5. Expected survival time > 3 months.
6. Presence of at least one measurable lesion according to RECIST 1.1 criteria.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-1.
8. Adequate organ function, with the following laboratory criteria:

   1. Absolute neutrophil count (ANC) ≥ 1.5x10^9/L, without the use of granulocyte-colony stimulating factor in the past 14 days.
   2. Platelet count ≥ 90x10^9/L, without transfusion in the past 14 days.
   3. Hemoglobin > 9 g/dL, without transfusion or use of erythropoietin-stimulating agents in the past 14 days.
   4. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN).
   5. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times ULN (ALT or AST ≤ 5 times ULN for patients with liver metastases).
   6. Serum creatinine ≤ 1.5 times ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 60 ml/min.
   7. Coagulation function within normal limits, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN.
   8. Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects with total triiodothyronine (T3) (or free T3) and free thyroxine (FT4) within the normal range can still be included.
   9. Normal cardiac enzymes (clinically insignificant isolated laboratory abnormalities are allowed, as determined by the investigator).
9. For premenopausal female subjects, a negative pregnancy test result (urine or serum) should be obtained within 3 days before the first dose of study drug (Day 1 of Cycle 1). If urine pregnancy test results cannot be confirmed as negative, a blood pregnancy test is required. Postmenopausal female is defined as at least 1 year after menopause or having undergone surgical sterilization or hysterectomy.
10. If there is a risk of pregnancy, all subjects (both male and female) must use contraception with a failure rate of less than 1% per year throughout the entire treatment period and for 120 days after the last dose of study drug.

Exclusion Criteria:

1. Diagnosis of malignant diseases other than extrahepatic bile duct cancer, excluding completely resected basal cell carcinoma, squamous cell carcinoma of the skin, and/or in situ carcinoma within the past 5 years.
2. Tumors located in the ampulla of Vater.
3. Currently participating in an interventional clinical study or received other investigational drugs or investigational device treatment within 4 weeks prior to the first dose of study drug.
4. Previously received therapy with anti-PD-1, anti-PD-L1, or anti-PD-L2 agents, or drugs targeting another T-cell receptor with inhibitory or co-stimulatory function (e.g., CTLA-4, OX-40, CD137).
5. Previously received palliative radiotherapy for biliary tumors, excluding postoperative adjuvant radiotherapy.
6. Received traditional Chinese medicine or immune modulatory drugs with anti-tumor indications within 2 weeks prior to the first dose of study drug (including thymosin, interferon, interleukins), except for local use to control pleural effusion.
7. Active autoimmune diseases requiring systemic treatment within 2 years prior to the first dose of study drug, or known history of primary immunodeficiency diseases. Patients with positive autoimmune antibodies alone will be evaluated by the investigator to determine if they have autoimmune diseases.
8. Currently receiving systemic corticosteroid therapy (excluding intranasal, inhaled, or topical corticosteroids) or any other form of immunosuppressive therapy within 4 weeks prior to the first dose of study drug. Physiological doses of corticosteroids (≤10 mg/day prednisone or equivalent) are permitted.
9. Uncontrolled pleural effusion or ascites that requires drainage or has not shown a significant increase in the past 3 days in patients who do not require drainage or whose drainage has been stopped.
10. Prior solid organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
11. Known hypersensitivity to the study drug, Candonilimab active substance, or excipients.
12. Insufficient recovery from any toxicities and/or complications related to previous interventions before starting treatment (i.e., ≤ Grade 1 or returning to baseline, excluding fatigue or alopecia).
13. Known history of human immunodeficiency virus (HIV) infection (i.e., positive for HIV 1/2 antibodies).
14. Untreated active hepatitis B defined as positive HBsAg and detectable HBV-DNA levels above the upper limit of normal at the study center. Note: The following HBV-infected patients may be included:

    HBV viral load <2.5 × 10^3 copies/mL (500 IU/mL) prior to the first dose of study drug, and patients should receive anti-HBV therapy throughout the study treatment.

    For patients who are anti-HBc positive, HBsAg negative, anti-HBs negative, and HBV DNA negative, no prophylactic anti-HBV therapy is required, but viral reactivation needs to be closely monitored.
15. Active hepatitis C infection (positive for hepatitis C virus (HCV) antibodies and HCV-RNA levels above the lower limit of detection).
16. Vaccination with live attenuated vaccines within 4 weeks prior to the first dose of study drug.
17. Pregnant or lactating women.
18. Presence of any severe or uncontrolled systemic diseases, including:

    Resting electrocardiogram with significant and symptomatic abnormalities in rhythm, conduction, or morphology, such as complete left bundle branch block, grade II or higher cardiac conduction block, ventricular arrhythmia, or atrial fibrillation.

    Unstable angina, congestive heart failure, chronic heart failure with New York Heart Association (NYHA) classification ≥ Grade 2.

    Any arterial thrombosis, embolism, or ischemia event within the past 6 months prior to enrollment, such as myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack.

    Major surgery (e.g., craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study drug or unhealed wounds, ulcers, or fractures. Minor surgical procedures, including venous puncture for intravenous infusion, within 7 days prior to the first dose of study drug are excluded.

    Poor blood pressure control (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg).

    Active pulmonary tuberculosis. Active or uncontrolled infections requiring systemic treatment. Clinical active diverticulitis, intra-abdominal abscess, or gastrointestinal obstruction.

    Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis.

    Poorly controlled diabetes (fasting blood glucose >10 mmol/L). Urine analysis showing urinary protein ≥++ and confirmed 24-hour urinary protein >1.0 g.

    Presence of psychiatric disorders that would hinder compliance with treatment.
19. Any medical history, evidence of disease, or abnormal laboratory values that could interfere with the study results, hinder the subject's full participation in the study, or pose other potential risks as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | through study completion, an average of 1 year
  Defined as the proportion of the subjects who have a complete response (CR) and partial response (PR) per RECIST 1.1 in enrolled subjects

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | through study completion, an average of 1 year

OTHER OUTCOMES:
overall survival (OS) | through study completion, an average of 1 year
  To evaluate the overall survival (OS) in order to assess the efficacy and safety of Candonilimab in combination with cisplatin and gemcitabine treatment.
progression free survival (PFS) | through study completion, an average of 1 year
  To evaluate the progression free survival (PFS) in order to assess the efficacy and safety of Candonilimab in combination with cisplatin and gemcitabine treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided